CLINICAL TRIAL: NCT01812434
Title: Evaluation of Phosphodiesterase-5 Inhibition on Endothelial Function in Heart Transplant Recipients
Brief Title: Phosphodiesterase-5 (PDE-5) Inhibition in Heart Transplant Recipients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left University
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1001M76094
Record Dates: First submitted 2012-02-20; First posted 2013-03-18 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Cardiac Allograft Vasculopathy
MeSH Terms: interventions — Sildenafil Citrate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Patients will be randomized to sildenafil arm taken three times a day for 28 days and then crossed over to the alternate arm.
  Interventions: Drug: Sildenafil
- Placebo (Experimental): Subject randomized to either Sildenafil or placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 20mg three time daily for 28 days
  Other Names: Viagra
  Arms: Sildenafil
Drug: Placebo — 20 mg three times daily for 28 days
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Hypothesis 1: Treatment of heart transplant recipients with sildenafil, a PDE-5 inhibitor, will improve small artery elasticity (SAE) when compared to placebo.

Hypothesis 2: PDE-5 inhibition will improve endothelial function, resulting in increased production of nitric oxide, reduced activation of circulating endothelial cells, and increased endothelial progenitor cells.

DETAILED DESCRIPTION:
Background and Significance In the United States, heart failure is an epidemic affecting 5,700,000 people, of which an estimated 100,000 to 200,000 suffer from end-stage heart failure. Cardiac transplantation has emerged as the definitive therapy for patients with end-stage heart failure.

Cardiac allograft vasculopathy (CAV) is the major limitation to longevity after heart transplant (HTx) and currently there are no effective treatments. It affects up to 45% of transplant recipients by year four post transplantation and is detectable on intravascular ultrasound in up to 75% at one year. Attempts to prevent cardiac allograft vasculopathy by modifying traditional risk factors such as dyslipidemia and hypertension have resulted in only modest improvements in outcomes after transplant. The efficacy of these preventive measures have been limited by the multifactorial nature of the process and the influence of nontraditional, less well-defined risk factors such as immune response, mode of brain death of the donor, and cytomegalovirus infection.

Both traditional and non-traditional risk factors do share a common final pathway, which is endothelial injury and subsequent endothelial dysfunction.

Endothelial dysfunction has been well described as a precursor to cardiac allograft vasculopathy in cardiac transplant recipients. While endothelial dysfunction is an integral part of the development of CAV and one of the earliest manifestations, it has not yet been demonstrated that targeting endothelial dysfunction delays or prevents the onset of cardiac allograft vasculopathy. Thus this study seeks to determine whether short-term sildenafil, when administered during the first 3 years after transplant, improves endothelial function in heart transplant recipients and thereby could prevent or delay cardiac allograft vasculopathy (CAV).

Rationale for using sildenafil Sildenafil has been demonstrated to dilate epicardial coronary arteries in patients with coronary artery disease and in those with normal coronary arteries who have risk factors for CAD and has been demonstrated to improve endothelial function in a variety of cardiovascular diseases including pulmonary hypertension and heart failure. By inhibiting PDE-5, an enzyme that metabolizes cyclic guanosine monophosphate (c-GMP), sildenafil enhances c-GMP-mediated relaxation and inhibits proliferation of vascular smooth-muscle cells. Inhibition of PDE-5 receptors with sildenafil appears to selectively improve endothelial function of the epicardial arteries; and in patients with severe CAD, sildenafil has been shown to improve coronary flow reserve. Based on these properties, we hypothesize that PDE-5 inhibition will improve endothelial function in transplant recipients and delay or prevent the onset of vasculopathy

Study Objectives

To determine the effect of Sildenafil on endothelial function in cardiac transplant recipients by:

1. Measuring the change in radial artery elasticity in HTx recipients before and after Sildenafil therapy.
2. Measuring change in number of endothelial progenitor cells before and after Sildenafil therapy

Study Design Overview of Study Design This is a randomized, double-blind, placebo-controlled 16 week crossover designed pilot study to evaluate the effect of oral sildenafil 20mg t.i.d, on small artery elasticity (SAE) and endothelial cells in heart transplant recipients.

Subjects will have pre-randomization and post treatment measurements of peripheral artery elasticity and endothelial progenitor cells Visits will occur at 0, 4, 8, 12 and 16 weeks. A graphic presentation of the study is shown below.

ELIGIBILITY:
Inclusion Criteria:

* Subject provided written informed consent
* Subject is 18 years old or Older
* Subject is a cardiac transplant recipient between 6 months - 5 years prior to week 0

Exclusion Criteria:

* Multi-organ transplant
* Been re-transplanted
* A contraindication to taking sildenafil
* Currently taking a PDE-5 inhibitor
* Mean arterial pressure < 65 mmHg
* A Left ventricular outflow obstruction
* A history or active retinitis pigmentosa
* Major surgery within 3 months of week 0
* Active infections to exclude are (CMV infection, febrile illness and Bacterial illness) within 3 months of week 0
* Acute rejection (grade 3A or greater) within 3 months of week 0
* Chronic kidney disease stage 4 (GFR<30 mL/min/1.73 m2) or acute renal failure
* Unstable cardiac disease, including myocardial infarction, stroke, or life- threatening arrhythmia within 6 months of week 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean change in SAE and in the number of endothelial progenitor cells after 4 weeks of treatment between placebo and sildenafil | 4 weeks
  Mean change in SAE after 4 weeks of treatment between placebo and sildenafil and mean change in the number of endothelial progenitor cells after 4 weeks of treatment

SECONDARY OUTCOMES:
Determine variability of SAE and large artery elasticity (LAE) in heart transplant recipients in order to plan a multi-center trial that will use arterial elasticity as a primary outcome | 16 weeks
  Mean change in SAE after 4 weeks of treatment between placebo and sildenafil and mean change in the number of endothelial progenitor cells after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Monica M Colvin-Adams, MD.MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States